CLINICAL TRIAL: NCT04453241
Title: A Randomized, Double-Blinded, Active Controlled, Phase I/ II Clinical Trial to Assess the Immunogenicity, Safety, and Tolerability of NBP615 Vaccine in Healthy Female Participants Aged 19 to 26 Years and Adolescent Aged 9 to 13 Years
Brief Title: Immunogenicity and Safety Study of NBP615 in Healthy Female
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SK Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-18062
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2020-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBP615 (Experimental): Adult : 3 doses of vaccination Adolescent :2 doses of vaccination
  Interventions: Biological: NBP615
- GARDASIL (Active Comparator): Adult : 3 doses of vaccination Adolescent :2 doses of vaccination
  Interventions: Biological: Gardasil

INTERVENTIONS:
Biological: NBP615 — Intramuscular injection, 0.5ml
  Arms: NBP615
Biological: Gardasil — Intramuscular injection, 0.5ml
  Arms: GARDASIL

SUMMARY:
This was a randomized, double-blind, active-controlled, phase I/II clinical trial to enroll 200 healthy female including 80 healthy adult aged 19 to 26 years and 120 adolescents aged 9 to 13 years.

DETAILED DESCRIPTION:
In order to confirm the safety, 80 healthy adult were enrolled first. Eligible subjects were randomized into 1:1 ratio to receive three doses of either test vaccine (NPB615) or comparator vaccine (Gardasil). The safety of the test vaccine (NBP615) was confirmed by 2nd vaccination in adult subjects. After that, enrolment of 120 adolescent subjects proceeded. Eligible subjects who previously agreed to participate in the study were screened and only those subjects who met the inclusion/exclusion criteria were randomized in to 1:1 to receive two doses of test vaccine (NBP615) or comparator (Gardasil pre-filled syringe). 0.5 ml Intramuscular injection at were given at each vaccination and two blood sample, pre vaccine and post vaccine 4 weeks after completion of vaccine were collected to assess the immunogenicity of NBP615 and Gardasil, comparator vaccine. Solicited adverse events occurred up to 7 days after each dose of the investigational product were collected in the diary card. Unsolicited adverse events occurred up to 28 days after each dose of the investigational product were collated in the diary card. Serious adverse events were collected during the entire study period. In addition to this safety data was collected through the study period by active contact with the study participants by doing home visit or by telephone contact.

ELIGIBILITY:
[Inclusion Criteria]

* Healthy adult(19 to 26 years)/adolescent(9 to 13 years) of age at the time of the 1st vaccination
* Participant fully understands study procedures, and voluntarily agrees to participate in the study and follow the study procedure by giving written informed consent

[Exclusion Criteria]

* Received a marketed Human papillomavirus(HPV) vaccine, or had participated in an HPV vaccine clinical trial and had received either active agent or placebo.
* History of hypersensitivity to any component of the study vaccines.
* Currently immunocompromised or was diagnosed as having a congenital or acquired immunodeficiency, Human Immunodeficiency Virus(HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease, other autoimmune condition, or other immune disorder which is decided to be medically significant by the investigator.
* Received immunoglobulins and/or blood product within 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Receiving or had received chemotherapy, immunosuppressive therapies, or radiation therapy in the year prior to enrolment.
* Chronic administration (>14 days) of immune-suppressants or immune modulating drugs within 3 months prior to the first vaccine dose or planned administration during the study period. Inhaled, nasal and topical steroids are allowed.
* Participant with severe thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections.
* Subject has active cervical disease or a significant history of cervical disease.

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2018-12-22 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer measured by Enzyme-linked Immunosorbent Assay(ELISA) | 4 weeks after the vaccination
  geometric mean titer against anti-HPV 6, 11, 16, and 18 for each treatment group
seroconversion rate measured by Enzyme-linked Immunosorbent Assay(ELISA) | 4 weeks after the vaccination
  proportion of subjects who seroconverted from seronegative at baseline to seropositive at post vaccination for anti-HPV 6, 11, 16, and 18
Geometric mean titer measured by pseudovirion-based neutralization assay(PBNA) | 4 weeks after the vaccination
  geometric mean titer against anti-HPV 6, 11, 16, and 18 for each treatment
Incidence rate of Solicited Adverse Event | 7 days after the vaccination
  Solicited local/systemic adverse event after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: k Zaman, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- SK Bioscience, Gyeonggi-do, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No